CLINICAL TRIAL: NCT03775187
Title: Expanded Access to Burosumab
Status: Available | Type: Expanded Access
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: UX023-EAP
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-09

CONDITIONS: X-linked Hypophosphatemia; Tumor-Induced Osteomalacia
Keywords: Expanded Access; Compassionate Use; XLH; TIO
MeSH Terms: conditions — Familial Hypophosphatemic Rickets; Oncogenic osteomalacia | interventions — burosumab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: Burosumab
  Other Names: UX023; Crysvita®; KRN23

SUMMARY:
Individual patient expanded access requests may be considered for patients who have no other treatment options

DETAILED DESCRIPTION:
Expanded access may be available outside of the US in countries prior to approval by the local regulatory agencies. For full details, please visit the links provided below.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult